CLINICAL TRIAL: NCT01068418
Title: Vitamin D Deficiency Augments Renin-Angiotensin System Activity in Obesity
Brief Title: Vitamin D Supplementation Reduces Renin-Angiotensin System Activity in Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jonathan S. Williams, MD, MMSc, Assistant Professor of Medicine, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2009p002062
Record Dates: First submitted 2010-02-11; First posted 2010-02-15 (Estimated); Results first posted 2017-02-14 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Obesity; Vitamin D Deficiency; Hypertension
Keywords: Obesity; Renin Angiotensin System; Vitamin D deficiency; Hypertension
MeSH Terms: conditions — Obesity; Vitamin D Deficiency; Hypertension | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitamin D3 (Experimental): 15000IU of vitamin D3 daily: open-label, single-arm
  Interventions: Dietary Supplement: Vitamin D (cholecalciferol)

INTERVENTIONS:
Dietary Supplement: Vitamin D (cholecalciferol) — cholecalciferol 15,000 IU daily for 30 days

SUMMARY:
Hypothesis: Vitamin D supplementation lower renin-angiotensin system activity in obesity.

Specific Aim: To investigate whether Vitamin D supplementation in obesity improves the vascular sensitivity to angiotensin II.

DETAILED DESCRIPTION:
Vitamin D deficiency and obesity are international epidemics that have both been associated with increased activity of the renin-angiotensin system (RAS). Because increased RAS activity is associated with cardiovascular disease, interventions to lower RAS will have favorable public health impacts.

This study aims to evaluate whether the supplementation of Vitamin D in obese subjects will lower local tissue RAS activity. RAS activity will be evaluated by cross-sectional measurement of RAS components and by quantifying the vascular response to an infusion of angiotensin II. Subjects will be studied while Vitamin D deficient, and will return for repeat study following Vitamin D supplementation, for comparison.

ELIGIBILITY:
Inclusion Criteria:

* age < 65,
* Cr < 1.6,
* 25-hydroxyvitamin D < 25 ng/mL,
* BMI > 30 kg/m2,
* stage I hypertension.

Exclusion Criteria:

* diabetes,
* coronary heart disease,
* heart failure,
* renal failure,
* liver failure,
* hyperparathyroidism,
* granulomatous disease.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2010-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S Williams, MD, MMSc, Principal Investigator — Brigham and Women's Hospital; Anand Vaidya, MD, Study Director — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin D3: This was a single-arm open-label study where participants received 15,000IU of vitamin D3 daily for 4 weeks.
Period: Overall Study
Arm/Group | Vitamin D3
Started | 26 (26 participants found to be eligible)
Medication Washout | 17 (9 participants were disempaneled during the medication washout phase due to noncompliance or high BP)
Completed | 14 (14 participants completed all study procedures.)
Not Completed | 12
Not completed — Physician Decision | 12

BASELINE CHARACTERISTICS:
Arm/Group | Vitamin D3
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14
Pre-Intervention Mean Arterial Pressure [Mean (Standard Deviation); unit: mmHg] | 105.6 (7.22)
Pre-Intervention 25-hydroxyvitamin D3 [Mean (Standard Deviation); unit: ng/mL] | 18.20 (6.76)
Pre-Intervention Parathyroid hormone concentration [Mean (Standard Deviation); unit: pg/mL] | 46.36 (16.09)
Pre-Intervention Serum calcium concentration [Mean (Standard Deviation); unit: mg/dL] | 8.94 (0.30)

OUTCOME MEASURES:

1. Primary Outcome: The Change in the Mean Arterial Blood Pressure in Response to an Infusion of Angiotensin II
Time Frame: baseline and 1 month following vitamin D3 therapy
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Vitamin D3
Number analyzed (Participants) | 14
mmHg | 1.97 (5.14)
Statistical Analysis 1: Comparison: Vitamin D3; A repeated measures regression analysis model was used to examine the effect of vitamin D3 therapy on the mean arterial pressure (mean of five measurements at each time point) before and during angiotensin II infusions, before and after vitamin D3 therapy; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis — Threshold for significance was P<0.05

2. Secondary Outcome: The Change in Renal Blood Flow in Response to an Infusion of Angiotensin II
Time Frame: baseline and 1 month following vitamin D3 therapy
Measure: Mean (Standard Deviation); unit: mL/min/1.72m2
Arm/Group | Vitamin D3
Number analyzed (Participants) | 14
mL/min/1.72m2 | -20.0 (40.7)
Statistical Analysis 1: Comparison: Vitamin D3; A repeated measures regression analysis model was used to examine the effect of vitamin D3 therapy on the renal plasma flow (mean of three measurements at each time point) before and during angiotensin II infusions, before and after vitamin D3 therapy; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis — threshold for significance was P<0.05

ADVERSE EVENTS:
Time Frame: 2.5 years
Arm/Group | Vitamin D3
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

LIMITATIONS AND CAVEATS:
This was a small physiologic study intended to provide insights on the influence of vitamin D3 on the renin-angiotensin system and vascular function. It is not generalizable to clinical practice. This is not a standard "clinical trial".

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No